CLINICAL TRIAL: NCT04705103
Title: Development of Artificial Intelligence Prediction Model for Uveitis Progression and Prognosis
Brief Title: Development of AI Model for Uveitis Progression and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Other Study IDs: 2020KYPJ185
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- initial
- relapse
- inactive

SUMMARY:
Uveitis is a recurrent inflammation of the eye that can lead to vision loss with various and complicated etiologies. There are many difficulties in uveitis management due to the requirement of long-term monitoring and treatment. This study intends to establish a longitudinal cohort of uveitis patients to colloect multimodal clinical data including visual acuity, intraocular pressure, anterior segment photography, fundus photography, fluoroscopy and other ophthalmic examinations, and final diagnosis in order to use artificial intelligence and deep learning technology to extract ocular features, explore the association with the progression and prognosis of uveitis and finally establish a disease management model for uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were diagnosed as uveitis, including the initial stage or relapse, or remission of uveitis.

Exclusion Criteria:

* Participants who cannnot cooperate with ocualr examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Initial stage of uveitis: The first episode of uveitis without treatment;
  2. Remission of uveitis: Uveitis caused by various reasons in the stable disease period of more than 3 months without treatment;
  3. Relapse of uveitis: After discontinuation of uveitis treatment, the disease stabilized for more than 3 months.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
uveitis progression | up to 1 month
  uveitis progression is divided into remission, relapse, or initial

IPD SHARING:
Plan to Share IPD: Undecided